CLINICAL TRIAL: NCT00663143
Title: Thiazolidinedione-Induced Bone Loss: Effects on Bone Marrow Stromal Cell Differentiation Capacity and Osteoblast Formation
Brief Title: Thiazolidinediones (TZD) Bone Loss and the Effects on Bone Marrow Differentiation and Osteoblast Formation
Acronym: TZDBONE
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Principal Investigator, Emory University
Other Study IDs: IRB00006692
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Osteoporosis
Keywords: investigate; TZD exposure; in vitro; alters; bone; formation; differentiation; capacity; bone marrow; stromal cells
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone Marrow
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stromal Cell Sample
  Interventions: Procedure: Stromal Cells Sample

INTERVENTIONS:
Procedure: Stromal Cells Sample — Human Bone Marrow Stromal Cells will be obtained from 5 patients. Stromal cells will be obtained from subjects undergoing bone graft procedure to repair traumatic mandible fractures. Bone graft specimens will be obtained from the ileac crest. This will allow easy access to bone marrow specimen without additional pain or complications. A total of 5 ml of bone marrow will be obtained from each patient.

SUMMARY:
Thiazolidinediones (TZDs) are a commonly used antidiabetic drugs currently used by over a million patients in the United States. Recent studies have shown that treatment with TZD may increase the risk of bone fractures. The cause of bone loss is not known. We believe that TZD may cause increased accumulation of fat in the bone marrow, which may cause decrease bone formation and weak bones. .

DETAILED DESCRIPTION:
This study aims to determine if TZDs increase the amount of fat and decrease the number of bone producing cells in the bone marrow.

A total of 5 subjects who require surgery for mandible (jaw) fracture and bone graft will be recruited. Some patients who will undergo mandible surgery will require a bone graft. In this procedure, a small piece of bone from the hip is placed in the mandible. In this study, a small amount of bone marrow fluid (5 mL or 1 teaspoon) will be obtained after the bone graft is completed. Obtaining the bone marrow will not result in additional pain or health problems. The effect of TZD on bone marrow and bone forming cells will be studied. The cells obtained during surgery will be grown at Dr Beck's laboratory at Emory University School of Medicine.

A working hypothesis suggests that the increased fracture risk in patients taking TZDs is the result of TZDs altering the differentiation capacity of bone marrow stromal cells pushing them towards the adipocyte lineage at the cost of osteoblast formation thereby decreasing bone formation.

Study AIM:To determine whether TZD exposure in vitro alters bone formation and the differentiation capacity of bone marrow stromal cells by promoting adipocyte lineage differentiation and lowering osteoblast formation.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years undergoing ileac crest bone graft to repair traumatic mandible fracture.
2. Patients admitted for elective or emergency surgery or trauma.

Exclusion Criteria:

1. Subjects with history of decompensated diabetes (blood glucose > 200 mg/dl)
2. Critically ill patients with multi-organ failure, relevant hepatic disease or impaired renal function (serum creatinine ≥ 2.0 mg/dl)
3. HIV
4. Hemolytic anemia and/or hematocrit < 28%
5. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
6. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with 1) traumatic mandibular (jaw) fracture who will undergo bone grafting or 2) trauma patients who will undergo intra-medullary rod placement for traumatic limb fractures will be considered as potential candidates in the study
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine whether TZD exposure in vitro alters bone formation and the differentiation capacity of bone marrow stromal cells by promoting adipocyte lineage differentiation and lowering osteoblast formation | once all subjects have been recruited

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia